CLINICAL TRIAL: NCT01328262
Title: A Randomized Clinical Trial on Hemoglobin Dose and Patient Matching
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Few patients, difficult to find suiting blood bags with the "right" weight.
Sponsor: Haukeland University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2010/476
Record Dates: First submitted 2011-02-24; First posted 2011-04-04 (Estimated); Results first posted 2025-04-17 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2019-02

CONDITIONS: Anemia
Keywords: Hemoglobins
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hemoglobin dose (Experimental): Intervention: Calculated red blood cell transfusion
  Interventions: Other: Calculated red blood cell transfusion
- Standard treatment (Active Comparator): Intervention: Standard red blood cell transfusion
  Interventions: Other: Standard red blood cell transfusion

INTERVENTIONS:
Other: Calculated red blood cell transfusion — The subjects receive an amount of red blood cells that has been calculated from their body surface area.
  Arms: Hemoglobin dose
Other: Standard red blood cell transfusion — The subjects in this group receive the prescribed number of red blood cell units.
  Arms: Standard treatment

SUMMARY:
The aim of this study is to evaluate whether the targeted hemoglobin increment (2 grams per decilitre) in the patient can be predicted from the hemoglobin dose/weight of the blood bag transfused. In the test group, the hemoglobin dose needed will be calculated, whereas in the control group, the prescribed number of red cell units will be transfused.

Hypothesis: By matching the hemoglobin dose to the individual needs of the patient the investigators will reduce the total usage of red cell concentrates.

DETAILED DESCRIPTION:
This is a randomized clinical study on hemoglobin dose and patient matching. The aim of the study is to evaluate whether the targeted hemoglobin increment (2 grams per decilitre) in the patient can be predicted from the hemoglobin dose/weight of the blood bag transfused. In the test group, the hemoglobin dose needed will be calculated, whereas in the control group, the prescribed number of red cell units will be transfused.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving red cell transfusions or expected to receive one or more red cell transfusions
* Patients over 16 years of age
* Patients for whom height and weight information is available
* Patients who have consented to participate

Exclusion Criteria:

* Patients who are hemodynamically unstable (ongoing bleeding or hemolysis)
* Patients with a known hemolytic anemia (congenital or acquired)
* Patients with a positive Direct Antiglobulin Test (DAT)
* Patients for whom informed consent has not been obtained
* Patients where the hemoglobin concentration increment target is above 2g/dl.
* Patients with auto- or alloantibodies against RBCs (red blood cells)..

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2010-11 (Actual); Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tor A Hervig, Professor, Principal Investigator
Locations (1):
- Haukeland University Hospital, Bergen, Norway

IPD SHARING:
Plan to Share IPD: No
If other scientists want to conduct a similar study, we will provide information that are completely anonymized. We are not in contact with any other research group now.

REFERENCES:
- [Derived] Radford M, Estcourt LJ, Sirotich E, Pitre T, Britto J, Watson M, Brunskill SJ, Fergusson DA, Doree C, Arnold DM. Restrictive versus liberal red blood cell transfusion strategies for people with haematological malignancies treated with intensive chemotherapy or radiotherapy, or both, with or without haematopoietic stem cell support. Cochrane Database Syst Rev. 2024 May 23;5(5):CD011305. doi: 10.1002/14651858.CD011305.pub3. PMID 38780066

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from November 2010 to January 2011 in the outpatient medical clinic at Haukeland University Hospital
Period: Overall Study
Arm/Group | Hemoglobin Dose | Standard Treatment
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Hemoglobin Dose | Standard Treatment | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Continuous [Mean (Full Range); unit: years] | 80 [70 to 89] | 76 [62 to 88] | 78 [62 to 89]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 5 | 4 | 9
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Norway | 6 | 6 | 12
Body Surface Area [Mean (Full Range); unit: m^2] | 1.81 [1.64 to 2.15] | 1.75 [1.52 to 2.01] | 1.78 [1.52 to 2.15]
Blood Volume [Mean (Full Range); unit: liter] | 4.7 [4.2 to 5.8] | 4.4 [3.3 to 5.4] | 4.6 [3.3 to 5.8]

OUTCOME MEASURES:

1. Primary Outcome: Hemoglobin Concentration Change
Description: The change in hemoglobin concentration after transfusion was recorded. The change is defined as hemoglobin (g/dl) after transfusion minus hemoglobin (g/dl) before transfusion.
Time Frame: Measurements of hemoglobin concentration taken from 30 min to 24hours after transfusion (earliest observation recorded)
Measure: Mean (Full Range); unit: g/dl
Groups:
- Hemoglobin Dose: Intervention: Calculated red blood cell transfusion
  Calculated red blood cell transfusion: The subjects receive an amount of red blood cells with a hemoglobin content that has been calculated from their body surface area.
Arm/Group | Hemoglobin Dose | Standard Treatment
Number analyzed (Participants) | 6 | 6
g/dl | 1.8 [1.2 to 2.3] | 2.0 [1.8 to 2.2]

ADVERSE EVENTS:
Time Frame: The adverse events were observed for 1 month after transfusion.
Groups:
- Hemoglobin Dose: Intervention: Calculated red blood cell transfusion
  Calculated red blood cell transfusion:
  The amount of hemoglobin needed to increase the patients' hemoglobin to the desired level is calculated based on their body surface area and blood volume. Blood bags are chosen by weight to match this amount of hemoglobin.
Arm/Group | Hemoglobin Dose | Standard Treatment
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/6 | 0/6

LIMITATIONS AND CAVEATS:
The study was terminated after just a couple of months as it proved to be hard to provide blood bags matching the desired amount of hemoglobin in the study group. This was further complicated by blood group alloantibodies in the patients restricting the choice of blood bags.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2010-11-01): https://cdn.clinicaltrials.gov/large-docs/62/NCT01328262/Prot_000.pdf